CLINICAL TRIAL: NCT03490110
Title: EEG Markers of Training-Induced Improvements in Cognitive Functioning
Brief Title: Brain Markers of Improvements in Cognitive Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N2240-P; 16-12-00774 (Other Grant/Funding Number: VA Northern California Health Care System)
Record Dates: First submitted 2017-11-09; First posted 2018-04-06 (Actual); Results first posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: TBI (Traumatic Brain Injury); Brain Injuries; Stress; Attention Deficit; Executive Dysfunction
Keywords: cognitive rehabilitation; EEG; TBI; brain networks; attention; memory; executive function
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: training in brain state regulation compared to treatment-as-usual
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- State regulation skill training (Experimental): This arm utilizes a training system designed to strengthen goal-directed cognitive-emotional state regulation skills. The emphasis is on practice and active application of skills across a range of challenge contexts. Digital scenarios provide experiential learning opportunities, allowing Veterans to apply skills to tackle challenges that are calibrated to maximize learning. Coaches guide learning for successful application of skills to challenges in personal life.
  Interventions: Behavioral: State regulation skill training
- Treatment-as-usual (Active Comparator): In this arm, participants receive clinical care as usual in VA and other clinics.
  Interventions: Other: Treatment-as-usual

INTERVENTIONS:
Behavioral: State regulation skill training — Participants complete seven supervised training sessions. Training sessions last 2 hours, and participants are requested to complete approximately 2.5 hours of additional skill practice over the course of each week outside of session (total ~4.5 hours per week).
  Arms: State regulation skill training
Other: Treatment-as-usual — Participants receive clinical care as usual over a matched time period.
  Arms: Treatment-as-usual

SUMMARY:
Some of the most common, persistent, and disabling consequences of traumatic brain injury affect an individual's ability to achieve personal goals. Interventions that strengthen abilities such as being able to concentrate, remember, stay calm and overcome challenges, could have far reaching benefits for Veterans. One challenge in rehabilitation is that response to training can be highly variable, and a better understanding of the neural bases for this variability could inform care. This pilot project will test the clinical behavioral effects of a cognitive skill training intervention and explore to what extent changes in markers of the brain's electrical activity (using the non-invasive technique of electroencephalograms, EEG) can explain differences in responses to skill training.

DETAILED DESCRIPTION:
Detailed Description: Traumatic brain injuries (TBI) can impair cognitive functioning long after the initial trauma. Some of the most common, persistent, and disabling consequences of traumatic brain injury are deficits in higher order cognitive functions that direct more basic processes based on an individual's goals. Symptoms such as distractibility and difficulty holding goal-relevant information in memory can affect achievement of personal and professional goals. These cognitive problems can be exacerbated by post-traumatic stress (PTS) symptoms, commonly observed in the Veteran population. Interventions that strengthen goal-directed regulation of cognitive-emotion states could have far reaching benefits for Veterans.

One challenge in rehabilitation is that response to training can be highly variable, and a better understanding of the neural bases for this variability could inform patient care. Investigators have developed a system for training neurocognitive skills that can be used in rehabilitation neuroscience studies to elucidate the neural bases of improvements in cognitive functioning. The training system is designed to help patients improve goal-directed brain state regulation, and preliminary work has investigated brain network parameters that may predict response to training. Electroencephalography (EEG) potentially provides easily accessible markers for the neural bases of improvements with training.

Objectives in this pilot study are to investigate the potential of EEG markers to: (1) explain differential responses to attention regulation training; and (2) predict responses to training.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* History of TBI (as defined by the American Congress of Rehabilitation Medicine and VA, with reported plausible mechanism of head injury, loss of consciousness with some period of posttraumatic alteration in cognition), in the chronic, stable phase of recovery (>6 months from injury)
* On stable psychoactive medications (> 30 days)
* Able and willing to participate in EEG, training and, assessments

Exclusion Criteria:

* Severely apathetic/abulic, aphasic, or other reasons for being unable or unwilling to participate with the training tasks
* Severe cognitive dysfunction
* History of neurodevelopmental abnormalities
* Ongoing illicit drug or alcohol abuse
* Schizophrenia
* Bipolar disorder
* History of other neurological disorders
* Current medical illnesses that may alter mental status or disrupt participation in the study
* Active psychotropic medication changes
* There will be no restriction in regard to gender, race, and socioeconomic status

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Chen, MD MA, Principal Investigator — VA Northern California Health Care System, Mather, CA
Locations (1):
- VA Northern California Health Care System, Mather, CA, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Started | 9 | 9
Completed | 6 | 6
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | State Regulation Skill Training | Treatment-as-usual | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (9.00) | 38.00 (9.61) | 39.29 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 8 | 9 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Composite Score of Attention and Executive Functioning From a Neurocognitive Test Battery
Description: The investigators created a composite score based upon standardized performance on the following neurocognitive measures of attention and executive functions: Wechsler Adult Intelligence Test - 4th Edition- letter number sequence; Auditory Consonant Trigrams - 9, 18, 36 second conditions; Digit Vigilance Test - Total Errors; Delis-Kaplan Executive Function System Color-Word Interference Trials 3 and 4 - Time and Total Errors; & Trails B - Time. Performance on each measure was scored using populations norms, and these scores are then standardized (Z-scored) and averaged to create a composite outcome (the unit measure being Z-score).
  A Z-score reflects the number of standard deviations a given score is away from the population mean: A Z-score of 0 is equal to the population mean, with positive and negative values reflecting performances above and below the population mean, respectively.
Time Frame: Week 1, before intervention period (baseline)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Number analyzed (Participants) | 6 | 6
units on a scale | 0.18 (0.79) | -0.06 (0.72)

2. Primary Outcome: Composite Score of Attention and Executive Functioning From a Neurocognitive Test Battery
Description: The investigators created a composite score based upon standardized performance on the following neurocognitive measures of attention and executive functions: Wechsler Adult Intelligence Test - 4th Edition- letter number sequence; Auditory Consonant Trigrams - 9, 18, 36 second conditions; Digit Vigilance Test - Total Errors; Delis-Kaplan Executive Function System Color-Word Interference Trials 3 and 4 - Time and Total Errors; & Trails B - Time. Performance on each measure was scored using populations norms, and these scores are then standardized (Z-scored) and averaged to create a composite outcome (the unit measure being Z-score).
  A Z-score reflects the number of standard deviations a given score is away from the population mean: A Z-score of 0 is equal to the population mean, with positive and negative values reflecting performances above and below the population mean, respectively.
  Change will be analyzed for this data as change from before to after the intervention period.
Time Frame: Week 8, after the intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Number analyzed (Participants) | 6 | 6
units on a scale | 0.49 (0.75) | -0.13 (0.45)

3. Secondary Outcome: Change in Event-Related Potential (ERP) Related to Memory Retrieval (Measured in uV)
Description: Electroencephalography (EEG) will be collected during tasks that require attention and working memory. The old/new ERP effect (difference between brain responses to correctly remembered studied items vs. correctly rejected unstudied items) will be analyzed for this data as change from before to after the intervention period.
Time Frame: Week 8, after the intervention period
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Number analyzed (Participants) | 6 | 6
uV
  EEG Electrode - Pz | 1.55 (1.88) | -0.42 (1.58)
  EEG Electrode - CPz | 2.27 (2.61) | 0.32 (1.17)

4. Secondary Outcome: Event-Related Potential (ERP) Related to Memory Retrieval (Measured in uV)
Description: Electroencephalography (EEG) will be collected during tasks that require attention and working memory. The old/new ERP effect (difference between brain responses to correctly remembered studied items vs. correctly rejected unstudied items) will be analyzed for this data prior to the intervention period.
Time Frame: Week 1, before the intervention period
Measure: Mean (Standard Deviation); unit: uV
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Number analyzed (Participants) | 6 | 6
uV
  EEG Electrode - Pz | 0.56 (1.06) | -0.07 (1.37)
  EEG Electrode - CPz | 1.41 (2.30) | 0.60 (0.99)

5. Secondary Outcome: Network Modularity From EEG
Description: EEG will be collected during a focused rest condition. Network modularity will be estimated from a matrix of connections between electrodes based on phase coherence, a unit-less measure of correlation between phase angles of EEG signals in the theta (4-8 Hz) frequency range. The modularity metric reflects the strength of modular network organization by summing the difference between the fraction of within-module connections to the total fraction of connections across modules, thus ranging from 0 (random) to 1 (completely modular). Change in network modularity will be analyzed for this data as change from before to after the intervention period.
Time Frame: Week 8, after the intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | State Regulation Skill Training | Treatment-as-usual
Number analyzed (Participants) | 6 | 6
units on a scale | 0.001 (0.018) | -0.002 (0.013)

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | State Regulation Skill Training | Treatment-as-usual
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT03490110/Prot_SAP_000.pdf